CLINICAL TRIAL: NCT00692328
Title: Expectation and Response to Levodopa & Acupuncture in Parkinson's Disease
Brief Title: Expectation and Response to Levodopa and Acupuncture in Parkinson's Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Oregon Health and Science University (Other)
Collaborators: National Center for Complementary and Integrative Health (NCCIH) (NIH)
Responsible Party: Principal Investigator, Barry S. Oken, MD, Oregon Health and Science University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: U19AT002656-02 (NIH); U19AT002656-02 (NIH); AT002656-02
Record Dates: First submitted 2008-06-04; First posted 2008-06-06 (Estimated); Last update posted 2015-05-05 (Estimated); Status verified 2015-05

CONDITIONS: Parkinson's Disease
Keywords: fatigue; TMS; MEP
MeSH Terms: conditions — Parkinson Disease; Fatigue | interventions — Levodopa; Acupuncture Therapy

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 1 (Active Comparator): The subjects will be told they receive levodopa or acupuncture.
  Interventions: Behavioral: Levodopa or acupuncture
- 2 (Placebo Comparator): The subjects will be told they receive placebo/sham levodopa or acupuncture.
  Interventions: Behavioral: Levodopa or acupuncture
- 3 (Experimental): The subjects will be told they have 50% chance of receiving real or placebo/sham levodopa or acupuncture.
  Interventions: Behavioral: Levodopa or acupuncture

INTERVENTIONS:
Behavioral: Levodopa or acupuncture — Comparison of subject expectancy of receiving levodopa or acupuncture.

SUMMARY:
To investigate how levodopa and acupuncture affect fatigue and muscle function in people who suffer from Parkinson's disease. Subjects may choose to participate in levodopa or acupuncture part, or both. Study procedures include an exercise protocol, transcranial magnetic stimulation (a non-invasive type of brain stimulation that cause small muscle twitch), a blood draw, and personality surveys.

DETAILED DESCRIPTION:
Subjects will answer surveys, have their blood drawn, undergo TMS and perform an exercise. The TMS/exercise task will measure fatigue and muscle response. The surveys will describe personality and measure fatigue. The CTRC will do genotype studies on the blood to look for genetic differences. Each subject is eligible to receive both study treatment types (levodopa and acupuncture). Depending upon the study treatment type they choose, each subject will be randomly assigned to one of six possible subject groups:

Ia. Full expectancy; levodopa: Subjects will be told that they are taking levodopa.

Ib. Half expectancy; levodopa: Subjects will be told that they have 50% chance of receiving levodopa or placebo.

Ic. No expectancy; levodopa: Subjects will be told that they are receiving placebo levodopa.

IIa. Full expectancy; acupuncture: Subjects will be told that they are receiving real acupuncture.

IIb. Half expectancy; acupuncture: Subjects will be told that they have 50% chance of receiving real or sham-acupuncture.

IIc. No expectancy; acupuncture: Subjects will be told that they are receiving sham-acupuncture.

Subjects will attend four visits for the levodopa part and/or three visits in the acupuncture part. On the first visit, subjects will answer questionnaires and have samples of their blood collected. On the other visits, subjects will undergo TMS while they perform a repetitive exercise task. Subjects will then either wait for 30 minutes or receive the investigative intervention that they have been randomly assigned for that particular visit, and then repeat the TMS/exercise task.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of Parkinson's disease
* Able to withdraw Parkinson's disease medication for 12 hours prior to a study visit
* Must be currently using levodopa to qualify for the levodopa part of the study

Exclusion Criteria:

* History of seizures
* Presence of any metal in the body, including DBS stimulators, pacemakers, metal plates or pins
* Severe cognitive deficits or psychosis
* Evidence of any clinically unstable disease, such as cancer, HIV/AIDS; unstable heart condition or other conditions that might require hospitalization
* Evidence of another neurological disease, such as multiple sclerosis, amyotrophic lateral sclerosis, or Huntington's disease

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 63 (Actual)
Dates: Start 2005-08; Primary Completion 2007-02 (Actual); Study Completion 2007-02 (Actual)

PRIMARY OUTCOMES:
Fatigue rate and muscle response evoked by transcranial muscle stimulation (TMS) | Before and immediately after the intervention

CONTACTS AND LOCATIONS:
Overall Officials: Jou-Shin Lou, MD, PhD, Principal Investigator — Oregon Health and Science University
Locations (1):
- Oregon Health & Science University, Portland, Oregon, United States